CLINICAL TRIAL: NCT02581059
Title: A Randomized Phase II Trial to Evaluate the Efficacy of Supportive Therapy With Ginseng for Patients on Treatment With Regorafenib
Brief Title: Efficacy of Ginseng for Patients on Regorafenib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder terminated.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Bayer (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00035502; HCRN GI14-191 (Other: Hoosier Cancer Research Network)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer; Palliative Medicine; Supportive Care
Keywords: Regorafenib; American Ginseng; Fatigue
MeSH Terms: conditions — Colorectal Neoplasms; Fatigue | interventions — regorafenib; Asian ginseng

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regorafenib + Ginseng (Experimental): Regorafenib will be administered 160 mg once daily for the first 21 days of each 28-day cycle. Subjects will receive 1,000 mg ginseng orally twice daily every day for 4 weeks (2 cycles).
  Interventions: Drug: Regorafenib; Dietary Supplement: Ginseng
- Regorafenib Only (Active Comparator): Regorafenib will be administered 160 mg once daily for the first 21 days of each 28-day cycle for 2 cycles.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — All subjects will receive regorafenib 160 mg orally once daily for the first 21 days of each 28-day cycle for 2 cycles.
  Other Names: Stivarga
Dietary Supplement: Ginseng — Subjects randomized to ginseng will receive 1,000 mg orally twice every day of each 28-day cycle for 2 cycles.
  Other Names: Panax quinquefolius
  Arms: Regorafenib + Ginseng

SUMMARY:
This is a randomized, multi-center phase II study of ginseng in colorectal cancer patients treated with regorafenib to determine if ginseng will reduce fatigue in this patient population and improve adherence to regorafenib. Ninety (90) subjects will be enrolled and randomized using a 2:1 allocation, with 60 subjects enrolled in the regorafenib + ginseng group and 30 enrolled in the regorafenib + no ginseng group.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

INVESTIGATIONAL TREATMENT:

Regorafenib will be administered 160 mg orally once daily for the first 21 days of each 28-day cycle. Subjects that randomize to receive ginseng will take 1,000 mg orally twice daily every day for 4 weeks (2 cycles). Subjects that randomize to NOT receive ginseng will not be given ginseng. Subjects will be instructed to take regorafenib with a low-fat meal.

Subjects will undergo fatigue assessments, using the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) instrument and Patient-Reported Outcomes Measurement Information System (PROMIS). Subjects will have a pill count cycle 2 day 1 (C2D1) and at the end of treatment visit. Subjects will have the re-staging scan (CT of chest/abdomen/pelvis) at the end of Cycle 2/ week 8 (±5).

Adequate bone marrow, liver and renal function assessed by the following laboratory values obtained within 7 days prior to registration for protocol therapy:

Hematopoietic:

* Absolute neutrophil count (ANC) count > 1,500/mm^3
* Hemoglobin (Hgb) > 9g/dL
* Platelet count > 100,000/mm^3

Renal:

* Serum creatinine ≤ 1.5 × the upper limit of normal (ULN)

Hepatic:

* Total bilirubin ≤ 1.5 × the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN (≤ 5 × ULN for subjects with liver involvement of their cancer)
* Alkaline phosphatase (ALP) limit ≤ 2.5 × ULN (≤ 5 × ULN for subjects with liver involvement of their cancer)

Coagulation:

* International normalized ratio (INR)/Partial thromboplastin time (PTT) ≤ 1.5 × ULN. NOTE: Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate if no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable, based on a measurement that is pre-dose as defined by the local standard of care. Warfarin does should not exceed 1 mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and be willing to sign the written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization for release of personal health information. A signed informed consent form (ICF) must be appropriately obtained prior to the conduct of any trial-specific procedure. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* Life expectancy of at least 12 weeks (3 months) as determined by the treating physician.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 28 days prior to registration.
* Histological or pathologically confirmed stage IV adenocarcinoma of the colon.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 2 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the treating physician or a designated associate. NOTE: Examples of adequate contraception may include but are not limited to a combination of any two of the following: use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods of contraception (condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/ film/cream/vaginal suppository); total abstinence; male/female sterilization
* All subjects must have radiographically assessable disease per RECIST v1.1 obtained by imaging within 28 days prior to registration.
* Must be able to swallow and retain oral medication.
* Subject must be deemed a suitable candidate for regorafenib as per their treating physician.

Exclusion Criteria:

* Subject should not be receiving any agent for fatigue including steroids, megace or opioids. NOTE: Subjects who have a contrast-induced allergy are allowed to receive steroids for their scans.
* Radiotherapy within 2 weeks prior to study registration. Subjects must have recovered from all therapy-related toxicities.
* Prior treatment with regorafenib.
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
* Congestive heart failure > New York Heart Association (NYHA) class 2: unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), myocardial infarction less than 6 months before study registration; cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted); uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to study registration.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months of study registration.
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 3 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (Non-invasive tumor), Tis (Carcinoma in situ) and T1 (Tumor invades lamina propria)].
* Subjects with pheochromocytoma.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2 NCI-CTCAE v4.0.
* Metastatic brain or meningeal tumors (symptomatic or asymptomatic).
* Major surgical procedure or significant traumatic injury, as defined by the site investigator, within 28 days before study registration.
* Renal failure requiring hemo- or peritoneal dialysis
* Dehydration Grade > 2 NCI CTCAE v4 within 7 days prior to registration.
* Subjects with seizure disorder currently requiring medication.
* Persistent proteinuria ≥ Grade 3 NCI CTCAE v4.0 as defined as > 3.5 g/24 hours, measured by urine protein: creatinine ratio on a random urine sample.
* Interstitial lung disease with ongoing signs and symptoms at the time of study registration.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI CTCAE version 4.0 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition which, in the opinion of the treating physician, will affect the absorption of any of the agents used in this study.
* Women who are pregnant or breast-feeding.
* Any condition, which, in the site investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Treatment with any investigational agent within 28 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodwige J. Desnoyers, M.D., Study Chair — Hoosier Cancer Research Network
Locations (5):
- United States (5):
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Altantic Health System, Morristown, New Jersey
  - Comprehensive Cancer Center at Wake Forest Baptist, Winston-Salem, North Carolina
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Study Treatment
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Started | 4 | 6
Completed | 0 | 1
Not Completed | 4 | 5
Not completed — Disease Progression | 1 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 1
Not completed — Patient Withdrawal After Therapy Start | 0 | 1
Not completed — Screen Failure Before Therapy Start | 0 | 1
Period: Follow up
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 3 | 5
Completed | 0 | 0
Not Completed | 3 | 5
Not completed — Death | 1 | 3
Not completed — study terminated | 1 | 1
Not completed — screen failure | 0 | 1
Not completed — Patient started new clinical trial | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib Only | Regorafenib + Ginseng | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic | 4 | 6 | 10
  Ethnicity: Hispanic | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG performance status :
  0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 0 | 1 | 1
    1 | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Subject Fatigue Assessment--Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF)
Description: MFSI-SF is a 30-item self-report instrument designed to measure general fatigue, physical fatigue, emotional fatigue, mental fatigue, and vigor--each scored on a 5-point Likert scale from 0 ("not at all") to 4 ("extremely"). The total score is calculated by adding the general, physical, emotional, and mental subscale scores and subtracting the vigor subscale score. Thus, total scores can range from -24 to 96 where higher scores indicate more of the cancer-related fatigue (meaning higher scores represent worse fatigue). A minimally clinically important improvement (or worsening) in the MFSI-Short Form is for changes of more than 4.5 points. T-score value of 36 indicates the population mean with a standard deviation of 34.93.
Time Frame: From date of first dose until end of cycle 2 (8 weeks)
Population: Data not collected for one in each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Number analyzed (Participants) | 3 | 4
score on a scale | 5.33 (8.39) | 8.50 (23.84)

2. Primary Outcome: Subject Fatigue Assessment--Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Each of the total raw scores were translated into T-scores for each participant using scoring tables for converting the PROMIS short form. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A higher PROMIS T-score represents more of the concept being measured. For this instrument all questions were negatively worded (i.e., How fatigued were you on average?) therefore a higher T-score represents having more fatigue. Thus, a T-score of 60 is one SD
Time Frame: From date of first dose until end of cycle 2 (8 weeks)
Population: Data not collected from one participant in each group.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Number analyzed (Participants) | 3 | 4
T-Score | 18 (6.24) | 22.75 (11.64)

3. Secondary Outcome: Subject Compliance
Description: Pill counts will be used to assess adherence to regorafenib and ginseng for subjects on each arm. Overall percentage reported.
Time Frame: Cycle 1 From date of first dose until day 15
Population: Data not collected from missing participants in each group/arm.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Groups:
- Regorafenib + Ginseng Arm (Regorafenib Compliance Only): Regorafenib compliance only for the Regorafenib + Ginseng Arm Regorafenib: All subjects will receive regorafenib 160 mg orally once daily for the first 21 days of each 28-day cycle for 2 cycles.
- Regorafenib + Ginseng Arm (Ginseng Compliance Only): Ginseng compliance for Regorafenib + Ginseng arm
  Ginseng: Subjects randomized to ginseng will receive 1,000 mg orally twice every day of each 28-day cycle for 2 cycles.
Arm/Group | Regorafenib Only | Regorafenib + Ginseng Arm (Regorafenib Compliance Only) | Regorafenib + Ginseng Arm (Ginseng Compliance Only)
Number analyzed (Participants) | 1 | 0 | 1
percentage of pills taken | 100 |  | 75

4. Secondary Outcome: Subject Compliance
Description: as for outcome 3
Time Frame: Cycle 2 From date of first dose until day 15
Population: Data was not collected from missing participants in each group/arm.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Arm/Group | Regorafenib Only | Regorafenib + Ginseng Arm (Regorafenib Compliance Only) | Regorafenib + Ginseng Arm (Ginseng Compliance Only)
Number analyzed (Participants) | 1 | 1 | 2
percentage of pills taken | 75 | 100 | 100 (50)

5. Secondary Outcome: Subject Compliance
Description: as for outcome 3
Time Frame: Cycle 1 From day16 until day 22
Population: Data was not collected from missing participants in each group/arm.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Arm/Group | Regorafenib Only | Regorafenib + Ginseng Arm (Regorafenib Compliance Only) | Regorafenib + Ginseng Arm (Ginseng Compliance Only)
Number analyzed (Participants) | 1 | 1 | 1
percentage of pills taken | 100 | 75 | 100

6. Secondary Outcome: Subject Compliance
Description: as for outcome 3
Time Frame: Cycle 2 From day 16 until day 22
Population: Data was not collected from missing participants in each group/arm.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Arm/Group | Regorafenib Only | Regorafenib + Ginseng Arm (Regorafenib Compliance Only) | Regorafenib + Ginseng Arm (Ginseng Compliance Only)
Number analyzed (Participants) | 1 | 0 | 1
percentage of pills taken | 75 |  | 50

7. Secondary Outcome: Characterize Adverse Events (AE)
Description: Toxicity assessed using Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0) criteria
Time Frame: From date of first dose until end of cycle 2 (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Number analyzed (Participants) | 4 | 6
Participants
  Acute Kidney Injury | 0 | 1
  ALANINE AMINOTRANSFERASE INCREASED | 0 | 1
  HEPATOBILIARY DISORDERS | 0 | 1

8. Secondary Outcome: Subject Retention
Description: Retention will be determined by the proportion of subjects on each arm who complete the study.
Time Frame: From date of first dose until end of cycle 2 (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Number analyzed (Participants) | 4 | 6
Participants
  Started | 4 | 6
  Completed (total retained number) | 0 | 1

9. Secondary Outcome: Evaluate Response Rate (RR)
Description: the number of subjects with confirmed partial response (PR) or complete response (CR) according to RECIST v.1.1, from the start of treatment until disease progression/recurrence
Time Frame: From cycle 1 day 1 (C1D1) until death or up to 18 months
Population: Data not collected for this outcome from missing participants in each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Overall Survival
Description: date of randomization to date of death from any cause
Time Frame: From C1D1 until death or up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
Number analyzed (Participants) | 4 | 6
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Begin C1D1 and every chemotherapy cycles (4 weeks) thereafter, for up to 18 months or until unacceptable toxicity.
Arm/Group | Regorafenib Only | Regorafenib + Ginseng
All-Cause Mortality (participants affected / at risk) | 2/4 | 4/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Only (N=4) | Regorafenib + Ginseng (N=6)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Only (N=4) | Regorafenib + Ginseng (N=6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 4 (6)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (3) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
EDEMA LIMBS (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 3 (7) | 4 (9)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (3) | 2 (5)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 1 (2)
MALAISE (General disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (6) | 2 (2)
RASH PUSTULAR (Infections and infestations) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (3)
WEIGHT LOSS (Investigations) | 3 (3) | 3 (5)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (3)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (9)
BLURRED VISION (Eye disorders) | 0 (0) | 1 (1)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 1 (2)
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1)
CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 3 (5)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (2)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
RECTAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT02581059/Prot_SAP_000.pdf